CLINICAL TRIAL: NCT06815367
Title: Comparing the Effects of Pneumatic Compression and Blood Flow Restriction Therapy on Muscle Recovery
Brief Title: Pneumatic Compression vs Blood Flow Restriction for Muscle Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Todd Schroeder, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-23-00594
Record Dates: First submitted 2024-09-17; First posted 2025-02-07 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Delayed Onset Muscle Soreness
MeSH Terms: interventions — Intermittent Pneumatic Compression Devices; Blood Flow Restriction Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): The participants will be asked to refrain from exercise 24 hours prior to and following the exercise. Participants will complete all pre-exercise tests (DOMS, CMJ, MVIC). The exercise consists of running on a treadmill situated at a -10% grade at 9 km/hr (5.59 mph) for 20 minutes. This is proceeded and followed by 5 minute warm-up/cool-down periods.
  Those that are allocated to the "control" group, will not receive treatment after the downhill running protocol.
- Pneumatic compression (Experimental): The participants will be asked to refrain from exercise 24 hours prior to and following the exercise. Participants will complete all pre-exercise tests (DOMS, CMJ, MVIC). The exercise consists of running on a treadmill situated at a -10% grade at 9 km/hr (5.59 mph) for 20 minutes. This is proceeded and followed by 5 minute warm-up/cool-down periods. Those allocated to the "pneumatic compression" group will receive 20 minutes of pneumatic compression at 100 mmHg.
  Interventions: Device: Pneumatic Compression
- Blood flow restriction (Experimental): The participants will be asked to refrain from exercise 24 hours prior to and following the exercise. Participants will complete all pre-exercise tests (DOMS, CMJ, MVIC). The exercise consists of running on a treadmill situated at a -10% grade at 9 km/hr (5.59 mph) for 20 minutes. This is proceeded and followed by 5 minute warm-up/cool-down periods.
  Those allocated to the "BFR" group will receive 4 rounds of treatment: 3 minutes will be spent at 100% of resting limb occlusion pressure, followed by 2 minutes of 0% occlusion.
  Interventions: Device: Blood Flow Restriction

INTERVENTIONS:
Device: Pneumatic Compression — Following downhill running protocol, participants will complete 20 minutes of pneumatic compression at 100 mmHg.
  Arms: Pneumatic compression
Device: Blood Flow Restriction — Following the downhill running protocol, participants will complete 4 rounds of treatment: 3 minutes at 100% resting limb occlusion pressure, 2 minutes of 0% resting limb occlusion pressure.
  Arms: Blood flow restriction

SUMMARY:
Both BFR and intermittent pneumatic compression are purported to decrease symptoms associated with exercise induced muscle damage (EIMD) that cause delayed onset muscle soreness (DOMS). Blood flow restriction relies on applying pressurized cuffs to the most proximal portion of the limb. Another form of recovery often relied upon is pneumatic compression. The mechanism by which pneumatic compression works is similar to that of a massage, whereby the device progressively increases the pressure on a portion of the limb before releasing and moving further up the limb.The purpose of this study is determine whether BFR or pneumatic compression can be used to decreased DOMS which may indicate enhanced recovery.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years of age
* Recreationally active population
* Women should be on a form of hormonal contraception.
* No current musculoskeletal injuries or pathologies
* Must answer "yes" to all PAR-Q questions.

Exclusion Criteria:

* Individuals that routinely train trail running
* Discomfort when running
* Deep vein thrombosis
* Blood clots
* Cancerous lesions
* Sensory or mental impairment
* Unstable fractures
* Acute pulmonary edema
* Acute thrombophlebitis
* Acute congestive cardiac failure
* Acute infections
* Episodes of pulmonary embolism
* Wounds, lesions, infection, or tumors
* Bone fractures or dislocations
* Increased venous and lymphatic return
* Answers "no" to any of the PAR-Q screening questions

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Counter Movement Jump Height | Immediately before and immediately after exercise, immediately after treatment, 24-hours post treatment.
  Participants will be asked to complete three consecutive counter movement jumps with hands on hips. The CMJ will be used as an indirect measure of muscle function.
Maximal Voluntary Isometric Contraction | Immediately before and immediately after exercise, immediately after treatment, 24-hours post treatment.
  Participants will be asked to complete an MVIC to assess muscle function.
Sedentary delayed onset muscle soreness | Immediately before and immediately after exercise, immediately after treatment, 24-hours post treatment.
  Using a visual analog scale, participants will be asked to rate their level of soreness while at rest.
Active delayed onset muscle soreness | Using a visual analog scale, participants will be asked to rate their level of soreness while at rest.
  Using a visual analog scale, participants will be asked to rate their level of soreness while completing a wall sit.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No